CLINICAL TRIAL: NCT04563624
Title: Clinical Assessment Accourding to Modified Usphs"of Indirect Restoration Fabricated From Nano Hybrid Composite Blocks Versus Ceramic Blocks in Badly Broken Teeth One Year Follow up Randomized Clinical Trial
Brief Title: Clinical Assessment of Indirect Restoration Fabricated From Nano Hybrid Composite Blocks Versus Ceramic Blocks in Badly Broken Teeth One Year Follow up
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haneen ahmed shafik elmoselhy, assistant lecturer in the operative department, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13919991
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Teeth Restoration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ceramic cad cam blocks (Experimental)
  Interventions: Drug: ceramic cad cam blocks
- composite cad cam blocks (Active Comparator)
  Interventions: Drug: composite blocks

INTERVENTIONS:
Drug: composite blocks — cad cam composite blocks
  Arms: composite cad cam blocks
Drug: ceramic cad cam blocks — ceramic cad cam blocks
  Arms: ceramic cad cam blocks

SUMMARY:
The aim of the study is to compare one-year clinical performance of indirect restoration fabricated from nano hybrid composite CAD CAM blocks and ceramic blocks

DETAILED DESCRIPTION:
This research is conducted for comparing the clinical efficacy of nano hybrid composite blocks and ceramic blocks ., the choice of nano hybrid composite blocks based on the claim of the manufacturer, as it's considered to be promising , nano hybrid composite blocks has the highest fillers content (86% by weight), resembles natural teeth perfectly , Excellent physical values for flexural strength and abrasion, No firing required (a real one step ), can be processed using any conventional milling unit, can be finished and polished optimally, Ideal for grinding even in cases with thin edges.

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly broken vital teeth
* Young adult Males or female
* Good oral hygiene measures
* Cooperative patients approving to participate in the study

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease
* Severe medical complications
* Lack of compliance
* Endodontically treated teeth

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
marginal integrity | one year
  using usphs visual inspection

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elmoselhy HAS, Hassanien OES, Haridy MF, Salam El Baz MAE, Saber S. Two-year clinical performance of indirect restorations fabricated from CAD/CAM nano hybrid composite versus lithium disilicate in mutilated vital teeth. A randomized controlled trial. BMC Oral Health. 2024 Jan 17;24(1):101. doi: 10.1186/s12903-023-03847-6. PMID 38233771